CLINICAL TRIAL: NCT03792815
Title: Open-labelled, Multicenter Phase II Clinical Trial of Intravenous Busulfan, Melphalan and Etoposide as Conditioning for Autologous Transplantation in Patients With Poor-risk, Refractory or Relapsed Non-Hodgkin's Lymphoma
Brief Title: Busulfan, Melphalan and Etoposide as Conditioning for Autologous Transplantation for Non-Hodgkin's Lymphoma (NHL)
Acronym: BME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong-Ho Won, professor, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH HMO
Record Dates: First submitted 2010-02-16; First posted 2019-01-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Transplantation Conditioning
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Busulfan; Melphalan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- busulfan melphalan etoposide (Experimental): busulfan 3.2 mg/kg/day i.v. on day -7, -6, and -5 etoposide 400 mg/m2 i.v. on day -5 and -4 melphalan 50mg/m2/day i.v. on day -3 and -2
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Etoposide

INTERVENTIONS:
Drug: Busulfan — busulfan 3.2mg/kg iv on day -8, -7, and -6,
  Other Names: Busulfex
Drug: Melphalan — melphalan 50mg/m2/day i.v. on day -3 and -2
  Other Names: Alkeran
Drug: Etoposide — etoposide 400 mg/m2 i.v. on day -5 and -4

SUMMARY:
The investigators developed a protocol utilizing once-daily intravenous busulfan/melphalan/etoposide regimen as a conditioning for high-dose therapy (HDT) in the patients with high risk or relapsed Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
Treatment:

busulfan 3.2 mg/kg/day i.v. on day -7, -6, and -5 etoposide 400 mg/m2 i.v. on day -5 and -4 melphalan 50mg/m2/day i.v. on day -3 and -2

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed aggressive NHL
2. Mantle cell lymphoma
3. salvage chemotherapy sensitive relapse/refractory NHL
4. Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2.
5. Age; 18-65
6. Adequate renal function: serum creatinine ≤ 1.5mg/dL
7. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value & Bilirubin < 2 X upper normal value

Exclusion criteria

1. low grade NHL
2. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
3. Other serious illness or medical conditions

   * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
   * History of significant neurological or psychiatric disorders
   * Active uncontrolled infection (viral, bacterial or fungal infection)
4. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
5. HIV (+)
6. Patients who have hepatitis B virus (HBV) (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
rate of event free survival | from date of ASCT until the the time of disease progression, relapse, or death, whichever came first, assessed at least 2 years
  calculate from the date of ASCT until the time of disease progression, relapse, or death

SECONDARY OUTCOMES:
rate of event free survival | at least 2 years
  calculate from the date of ASCT until the time of death from any causes
rate of regimen related toxicity | up to 6 months
  calculate toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Won, Professor, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided